CLINICAL TRIAL: NCT04307771
Title: Effectiveness of Smart-phone App in Improving Oral-Health Knowledge & Practices Among School Going Adolescents: A Randomized Control Trial
Brief Title: Effectiveness of Smart Phone Application in Improving Oral Health Behaviours of Adolescents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr.Javeria Nafis, Post Graduate Student, Department of Community Health Sciences, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 3539
Record Dates: First submitted 2020-03-11; First posted 2020-03-13 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Oral Hygiene

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- m-health application (Experimental): a mobile app designed to send reminders for brushing and give information on maintaining oral health
  Interventions: Behavioral: m-Health application
- Leaflet (Other): This is the control arm. An educational leaflet for maintaining oral hygiene will be given to participants in this arm
  Interventions: Behavioral: m-Health application

INTERVENTIONS:
Behavioral: m-Health application — Dental Buddy is a mobile application that has been designed to improve oral hygiene maintenance behaviours in teenagers
  Other Names: Dental Buddy

SUMMARY:
This study would be a first step towards mobile-health associated Sustainable Development Goals by World Health Organization, as there are no mobile-health driven oral health activities in Karachi, Pakistan. Concurrently, it will help in improving knowledge and practices of adolescents towards general dental hygiene as this age is crucial for the prognosis of newly erupted permanent teeth. This would help in preventing chronic problems of adulthood. This will also help in reducing the number of days missed from school, increasing self-confidence of individuals as bad breath has a negative impact on one's self-esteem and confidence, giving a positive sense of aesthetics and will also keep in check over-all body health.Persistent unmaintained dental hygiene also overburdens families due to its high-maintenance outcomes like caries and early tooth loss. Dental treatment is considered as fourth most expensive treatment in developing countries . According to recent studies, households of low and middle income countries are at a higher risk of falling below the poverty line due to expenditure on dental problems. Such a simple intervention making use of modern-day technology would enable adolescents to keep their oral health in check and would prevent them from facing consequences of poor oral health.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent of age between 14-19 years
* Having access to an android device at home; either personal or parents'
* Would be able to use the app twice every day- Having access to Wi-Fi at home- for downloading the app.
* Willing to give consent
* participate in the study till the follow-up period.

Exclusion Criteria:

* - Having mixed dentition
* Undergoing orthodontic treatment
* Should have no serious existing gingival or dental problems* that could hinder calculation of plaque or gingival scores
* Should have no serious existing gingival or dental problems* that could hinder routine brushing.
* Taking medications that have effect on gingival/dental health
* Having intrinsic or extrinsic enamel defects/ tooth malformations
* Having more than 1/3rd of the tooth stained due to areca nut chewing, smokeless tobacco (gutkha) chewing or cigarette smoking.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 152 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-03 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge scores | 6 weeks
  Knowledge scores will be assessed by a self-administered questionnaire with maximum score of 30 and minimum of 0. Higher scores mean better knowledge.
Practice scores | 6 weeks
  reduction in plaque index scores. score range 0-6. score 0 being the best and score 6 being the worst. Gingival index scores ranging from 0-6, score ) lesser (0) being the best and 6 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Shafquat Rozi, Dr, Study Director — Aga Khan University

IPD SHARING:
Plan to Share IPD: No